CLINICAL TRIAL: NCT04447898
Title: A Randomized, Double-blind, Placebo-controlled, Dose Escalation Phase I Study Assessing the Safety and Immune Response of PPV-06 Vaccine in Patient With Inflammatory Knee Osteoarthritis (KOA)
Brief Title: Dose Escalation Study Assessing the Safety and Immune Response of PPV-06 Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peptinov SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PPV06-01
Record Dates: First submitted 2020-05-04; First posted 2020-06-25 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose (Experimental): 10 μg + Montanide™ ISA 51 VG
  Interventions: Drug: PPV-06 10 μg; Drug: Placebo
- High dose (Experimental): 50 μg + Montanide™ ISA 51 VG
  Interventions: Drug: PPV-06 50 μg; Drug: Placebo

INTERVENTIONS:
Drug: PPV-06 10 μg — Low dose + Montanide™ ISA 51 VG in SC administration = 3 injections on Day 0, Day 28, and Day 112
  Arms: Low dose
Drug: PPV-06 50 μg — High dose+ Montanide™ ISA 51 VG in SC administration = 3 injections on Day 0, Day 28, and Day 112
  Arms: High dose
Drug: Placebo — Placebo+ Montanide™ ISA 51 VG in SC administration = 3 injections on Day 0, Day 28, and Day 112

SUMMARY:
PPV-06 immunotherapy targets interleukin-6 (IL-6), a key molecule of the immune system whose overproduction is implicated in many inflammatory and autoimmune diseases such as rheumatoid arthritis and osteoarthritis. The benefit of vaccination with PPV-06 is to induce, in response to immunizations, the production of antibodies directed against IL-6. The antibodies produced will neutralize the biological activity of IL-6 involved in the body's inflammatory process.

The primary objective is to evaluate the safety/tolerability of vaccination with PPV-06.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged over 40 years;
2. Diagnosis of primary inflammatory Knee Osteoarthritis (KOA),
3. Body mass index (BMI) of 18-32 kg/m2 at screening;
4. Patients with normal organ function at baseline
5. Contraceptives measures
6. In the investigator's opinion, the patient is capable and willing to comply with the requirements of the study;
7. Willing and able to sign a written informed consent;
8. Affiliated to social security insurance.

Exclusion Criteria:

1. Systemic Autoimmune or immunodeficiency disease;
2. Administration of non-steroidal anti-inflammatory drug (NSAID):
3. Administration of prednisone or having intra-articular corticosteroid injection or bolus intramuscular or intravenous treatment with corticosteroids;
4. Patients treated with biologics such as anti-TNFAlpha, anti-IL-6 and anti-CD-20
5. Participation in another investigational drug or vaccine trial;
6. Knee surgery planned before screening and throughout the study;
7. Knee surgery within the year of baseline;
8. Knee trauma within 2 months of baseline;
9. Chronic hepatitis B and/or C infection. Patients with previous infection, resolved in the past, are eligible;
10. HIV-positivity;
11. History of allergic reaction to any constituents of the study drug;
12. Diagnosis or history of any inflammatory arthritis;
13. Neurologic disorders involving the lower limbs;
14. History of malignancy within the last 5 years;
15. Uncontrolled congestive heart failure or hypertension, unstable heart disease
16. Evidence of any clinically significant abnormality on a chest X-ray which, in the opinion of the investigator, could represent active infection or latent tuberculosis;
17. Moderate or severe acute illness/infection, persistent diarrhea or vomiting on the day of vaccination;
18. Received any licensed, non-live vaccine within the 14 days before receipt of any dose of the study vaccine or is scheduled to receive any licensed, non-live vaccine within 30 days following receipt of any dose of the study vaccine;
19. Receipt of immune globulins, blood or blood-derived products;
20. Pregnant or lactating females;
21. The investigator considers the patient unfit for the study as a result of the medical interview, physical examination, or screening investigations.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with DLT defined as grade 3 or higher treatment-related adverse events (monitored in all patients during the study treatment until the End of Study (Week 42) or early termination). | From Baseline to Week 42 (End of Study)
  The primary outcome measure of this study is to evaluate the safety/tolerability of PPV-06 vaccination

SECONDARY OUTCOMES:
The occurrence of all adverse events (AEs) and serious adverse events (SAEs), including clinically significant abnormal haematological and biochemical values (monitored during the entire study period until End of Study (Week 42) or early termination). | From Baseline to Week 42 (End of Study)
  This secondary outcome measure of this study is to evaluate additional indicators of safety / tolerability
The quantification of inflammatory markers will be assessed at Baseline, W4, W12, W16, W24, W32 and End of Study (Week 42) or early termination by measuring IL-6, hsCRP and CRPM level in blood | From Baseline to Week 42 (End of Study)
  This secondary outcome measure of this study is to evaluate additional indicators of safety / tolerability
The quantification of Anti-IL-6 antibody production, isotypes characterization and anti-CRM197 antibody level in serum at Baseline, W4, W12, W16, W24, W32 and EoS or early termination | From Baseline to Week 42 (End of Study)
  This secondary outcome measure of this study is to evaluate the humoral immune response of PPV-06
The quantification of Anti-IL-6 neutralizing antibody level in vitro at W4, W12, W16, W24, W32 and EoS or early termination | From Baseline to Week 42 (End of Study)
  This secondary outcome measure of this study is to evaluate the humoral immune response of PPV-06
The quantification of specific T cell response and polarization (Th1, Th2 and Th17) assessed by IFNg, IL-5 and IL-17 Elispot assay at Baseline, W24, W32 or early termination. | From Baseline to Week 42 (End of Study)
  This secondary outcome measure of this study is to evaluate the cellular immune response of PPV-06
The quantification of proliferative CD4+T cells assessed by flow cytometry at Baseline, W24, W32 or early termination. | From Baseline to Week 42 (End of Study)
  This secondary outcome measure of this study is to evaluate the cellular immune response of PPV-06
The frequency of hIL-6 epitope-specific memory B cells assessed by ELISPOT assay, at Baseline, W24, W32 or early termination. | From Baseline to Week 42 (End of Study)
  This secondary outcome measure of this study is to evaluate the cellular immune response of PPV-06

CONTACTS AND LOCATIONS:
Locations (1):
- Cic Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided